CLINICAL TRIAL: NCT00606203
Title: Dose Milnacipran Prevent Depressive Symptoms in Patients With Acute Stroke?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Centapharm Inc Flory Co Ltd, Centapharm Inc Flory Co Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 96-0083
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Ischemic Stroke; Depression
MeSH Terms: conditions — Ischemic Stroke; Depression | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The aims of this study are to investigate the prophylactic effect of milnacipran in post stroke depression.
  Interventions: Drug: milnacipran
- B (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: milnacipran — taking milnacipran(50) 1#bid after stoke to prevent the occurence of depression
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
Depression is one of the important psychiatric sequelae after stroke. The prevalence of post stroke depression (PSD) is approximately 20-40%. Depression comorbid with stroke has been found to be associated with increased disability, cognitive function decline, poorer rehabilitation outcome and higher mortality rate.We are going to conduct a trial of prevention of psot stroke depression by prescribing milnacipran in advance.

DETAILED DESCRIPTION:
First visit (visit 0) will be performed in the first three days after patient is admitted to the neurological ward due to ischemic stroke. The purposes of the initial assessment include demographic data collection (age, gender, stroke location), initial interview to exclude past history of depression, substance abuse or psychosis. In addition, Ham-D, CGI, NIHSS, Barthel index, MMSE (please refer to the "instruments" listed below) are performed in the first visit. Patients whose MMSE<15 or Ham-D>10 will be excluded.

After being enrolled, patients stratified with stroke locations are randomized assigned to two groups: group A (treatment group with active antidepressant) or group B (placebo group). Variables such as age, gender, severity of the NIHSS, MMSE and Ham-D will be controlled during assignment and the cytokine level will be checked also as baseline. The cytokine that will be checked includes IL-1, IL-6, TNF-α,IFN-γ that were considered pro-inflammatory cytokine. The anti-inflammatory cytokine of IL-4 ,IL-10 and TGF-β will be checked also .Patients in group A will take Milnacipran (50mg) 1# QD from the first day of being enrolled into the study and will titrate to 1# BID one week later. Patients in both groups will be followed at 1st, 3rd, 6th, 9th, and 12th month after stroke. The Ham-D, TDQ, NIHSS, Barthel index, CGI, MMSE and cytokines will be assessed in each of the check point. Patients in either group A or group B will be withdrawn from the study and referred to psychiatric clinics for further alternative management if they developed depression (Ham-D>17). Cytokine levels in depressed patients will be compared with the randomly selected controlled group. All the interviewers are blinded to the patient's medication. If patients drop out, the reason will be clarified and recorded. Patients who suffered from recurrent stroke during study period still keep the same protocol that are followed continuously for one year unless patients request for withdrawal

ELIGIBILITY:
Inclusion Criteria:

* Consecutive admission due to first or recurrent ischemic stroke (image proved) and stroke occurred in preceding 4 weeks before admission. The onset of stroke was defined as the occurrence of abnormal neurological symptoms according to the patients' statement. The following period is 12 months after being included (for the first and third study aims), and follow for another 24 months to study the immunological aspect of PSD (for the second study aim).

Exclusion Criteria:

* TIA (transit ischemic attack)
* Impairment of communication or cognitive function (MMSE<15)
* Past history of depression, psychosis, severe substance abuse
* Taking antidepressants at least 2 weeks prior to stroke
* Concurrent possible depression (Ham-D>10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression rating scale | 0,1,3,6,9,12th

SECONDARY OUTCOMES:
Taiwanese depression questionnaire, quality of life, london handicap scale | 0,1,3,6,9,12th month

CONTACTS AND LOCATIONS:
Overall Officials: Hin-Yeung Tsang, MD,PHD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan